CLINICAL TRIAL: NCT00587028
Title: Cathartic-Free Dual Energy Computerized Tomography (DECT) Colonography.
Brief Title: Cathartic-Free DECT Colonography for Detection of Colonic Polyps
Status: Terminated | Type: Observational
Why Stopped: Administrative closed due to funding
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeff Fidler, Principal Investigator, Mayo Clinic
Other Study IDs: 981-05; R21CA110390 (NIH)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Colonic Polyps
Keywords: Colonography; Colonoscopy; Virtual; Computed Tomographic Colonography; Large intestine; colon
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Oral Omnipaque MCA: Ten participant minimum: for stool tagging two days preceding the CT colonography, if applicable, with oral Omnipaque. This cohort at Scottsdale Mayo Clinic only.
- IV Iodine MCR: Ten participant minimum: for intravenous iodine contrast dye. This cohort at Rochester Mayo Clinic only.
- NO oral and no IV MCR: Five participant minimum for no oral or IV contrast.
- Replacement Group: Five participant minimum for either cohorts 1, 2, or 3 as above should there be poor imaging results. A like prepped participant will replace that who had poor quality imaging to meet 25 imaging data sets.

SUMMARY:
Asses the clinical performance of dual-energy CTC for the detection of larger polyps 1 cm or larger without cathartic preparation.

DETAILED DESCRIPTION:
Determine the feasibility to differentiate polyps from stool with or without the use of contrast agents and to assess the feasibility and accuracy of dual energy techniques in a pilot patient study.

1.1 Formulate algorithms that use dual-energy information to quantitatively measure specific material density of colon polyps in physics based simulation.

1.2 Determine optimal scanning parameters on prototype CT equipment.

2.1 Measure the material composition density and Hounsfield number of polyps with and without simulated contrast enhancement.

2.2 Measure the accuracy of dual-energy techniques to differentiate between polyps and stool and if needed using a combination of simulated intravenous enhanced polyps and contrast material tagged stool.

3.0 Asses the clinical performance of dual-energy CTC for the detection of larger polyps 1 cm or larger without cathartic preparation.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a known colorectal polyp or colon carcinoma with pathology, at or greater than 1 cm in size on a colonoscopy that is completed either eight weeks before or after CT Colonography study visit.
* If receiving iodine oral or IV contrast, must have a creatinine less than 1.4 on record within last 30 days of study visit date. If no creatinine is available, one will be drawn for enrollment criteria purposes.

Exclusion Criteria:

* Pregnant females.
* Presence of colostomy or right hemicolectomy.
* Inflammatory bowel disease (Crohn's, chronic ulcerative colitis).
* Familial polyposis syndrome.
* Pregnant female.
* Creatinine at or greater than 1.4
* Severe or uncontrolled chronic obstructive pulmonary disease (COPD) or chronic obstructive lung disease (COLD).
* Iodine contrast allergy.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic, Rochester, Minnesota and Mayo Clinic, Scottsdale, Arizona Colonoscopy schedules.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Clinical performance of dual-energy CT colonography (CTC). | Three Months
  Detection of polyps in cathartic-free CTC using optimized dual-energy techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff L. Fidler, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No